CLINICAL TRIAL: NCT05815875
Title: The Effect of The STEADI Program on Falls and Falls Prevention in Neurosurgical Patients in Jordan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jehad Rababah, Associate Professor, King Abdullah University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 92-2023
Record Dates: First submitted 2023-03-17; First posted 2023-04-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Fall Patients
Keywords: Falls prevention; Neurosurgery patients; STEADI

STUDY DESIGN:
Intervention Model Description: This study will be conducted using a 1-month prospective quasi-experimental design.
  The study sample will be 70 neurosurgical patients at King Abdullah University Hospital. The study sample will be non-randomly divided into a control group (35 patients) and an intervention group (35 patients).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The STEADI program will be applied to this group of participants. The STEADI involves frequent assessment of patients' risk for falls and making appropriate changes to decrease the risk for falls.
  Interventions: Combination Product: STEADI Program
- Control (Active Comparator): The STEADI program will not be applied to the control group participants. This group will receive the usual care provided to the patients in the hospital.
  Interventions: Other: Routine care

INTERVENTIONS:
Combination Product: STEADI Program — The investigators will conduct STEADI Algorithm for Falls Prevention educational sessions for healthcare providers in the neurosurgery unit, including doctors, nurses, physical therapists, and pharmacists. All healthcare providers in the neurosurgery unit will be invited to attend the educational sessions. Their participation will be voluntary and no obligations will be made, though. Healthcare providers will be invited to attend one 2-hour educational session. In each session, The investigators will have between 8-10 healthcare providers. The educational sessions will be delivered in the classroom available in the neurosurgery unit to facilitate the healthcare providers' access. PowerPoint presentations, videos, quizzes, case studies, and in-class discussions will be used to deliver learning content during the educational sessions. Healthcare providers will then be asked to apply the STEADI interventions on a group of patients.
  Arms: Intervention
Other: Routine care — The control group participants will receive routine care. Routine care involves only assessing for falls using Morse Falls Scale (MFS). MFS assesses a patient's fall risk upon admission, following a change in status, and at discharge or transfer to a new setting.
  Arms: Control

SUMMARY:
The goal of this interventional study will be to evaluate the effectiveness of the STEADI Program on falls and falling prevention compared with routine falling assessment in neurosurgical patients in Jordan. The researchers will compare the effectiveness of the STEADI intervention in the intervention group. Participants in the intervention group will be assessed for falls risk using well-established tools as recommended by the Centers for Disease Control and Prevention (CDC). The control group participants will receive regular falling assessment which involves using Morse Fall Scale.

DETAILED DESCRIPTION:
The STEADI (Stopping Elderly Accidents, Deaths & Injuries) program was developed by the Centers for Disease Control and Prevention (CDC) to help healthcare providers address falls among older adults. The STEADI program provides healthcare providers with tools and resources to screen their older patients for fall risk, assess risk factors, and develop and implement an individualized fall prevention plan. The STEADI program is an evidence-based approach to fall prevention and has been shown to reduce falls among older adults. However, evidence regarding the effectiveness and usefulness of the STEADI among neurosurgery patients is lacking. The investigators of the current research will conduct a 2-hour educational session to train healthcare providers in a neurosurgery unit on using the STEADI tools and algorithm. Then, the investigators will collect data to assess whether applying the STEADI decreases the risk for falls in neurosurgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted patients to the neurosurgery unit as a case of neurosurgery, have ≥4 scores on the Stay Independent Brochure (SIB), 18 years old or older.

Exclusion Criteria:

* Bedridden and unconscious/comatose patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The Stay Independent Brochure (SIB) | Change from baseline to 5-days and 1-month
  The Stay Independent Brochure (SIB) will be used to assess the risk for falls as recommended by the CDC's STEADI. The SIB involves 12 items, and each item has a potential response of "No" (= 0) or "Yes" (= 1). Scoring relies on the number of "yes" answers to each question item, with a total possible score of 12. Participants are considered to be at risk of fall based on the following criteria: answer "yes" to 4 or more out of 12 questions, otherwise not at risk.
The clinician's 3 key questions | Change from baseline to 5-days and 1-month
  The clinician's 3 key questions will also be used to assess the risk for falls as recommended by the CDC's STEADI. The three questions used are "fell in the past year?" "feel unsteady when standing or walking?" and "worries about walking?" Participants with a "yes" answer to any of the 3 key questions will be considered at risk of falls, and those with all "no" answers will be considered not at risk for falls.
Time Up and Go (TUG) | Change from baseline to 5-days and 1-month
  The TUG is designed to evaluate mobility skills, balance, and fall risk. TUG performance is measured as the time taken to complete the test, with a longer completion time indicating poorer functional mobility and higher fall risk.
30-Second Chair Stand | Change from baseline to 5-days and 1-month
  The 30-S Chair Stand assesses lower extremity strength and endurance. This test uses a chair with a straight back without armrests and a seat height of 17 inches. The participant will sit in a chair with their arms crossed over their chest. When the investigator says "go," the participant will stand up and sit down again. And repeat this for 30 seconds. The investigator will count how many times a participant can do this. A lower number may mean the participant is at higher risk for a fall.
The 4-Stage Balance test | Change from baseline to 5-days and 1-month
  The 4-Stage Balance test is an assessment of static balance in four different positions and increasingly challenging positions: (1) feet together, (2) instep of foot advanced to toe of other foot, (3) foot in front of other foot (tandem), and (4) and single-leg stance. Without being able to stand or lasting less than 10 seconds, all 4 types are considered to be at risk for falls, standing for 10 seconds or more is considered not at risk for falls.
Actual falls | At final (1-month) assessment
  The actual number of falls will be recorded for all patients. Results will be reported as an average number of falls.

CONTACTS AND LOCATIONS:
Locations (1):
- Jehad Rababah, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers. Only aggregate data will be disseminated.

REFERENCES:
- [Result] Stevens JA, Phelan EA. Development of STEADI: a fall prevention resource for health care providers. Health Promot Pract. 2013 Sep;14(5):706-14. doi: 10.1177/1524839912463576. Epub 2012 Nov 16. PMID 23159993
- See also: This is the official link to the CDC's STEADI website — https://www.cdc.gov/steadi/index.html